CLINICAL TRIAL: NCT05930418
Title: Cardiovascular Magnetic Resonance Prognosticators In Pediatric Oncology Patients With Sepsis: A Priority Pilot Study
Brief Title: Cardiovascular Magnetic Resonance Prognosticators in Pediatric Oncology Patients With Sepsis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CRIMSON2; NCI-2023-04528 (Other: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2023-06-08; First posted 2023-07-05 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Acute Respiratory Distress Syndrome; Sepsis; Cardiovascular Shock
MeSH Terms: conditions — Respiratory Distress Syndrome; Sepsis; Shock, Cardiogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Cardiac MRI after sepsis (Experimental): Participants who meet the eligibility criteria of severe sepsis.
  Interventions: Diagnostic Test: Cardiac MRI

INTERVENTIONS:
Diagnostic Test: Cardiac MRI — Cardiac Magnetic Resonance provides more sensitive measure of ventricular volume and ejection fraction as well as novel markers of tissue characterization and edema assessment.

SUMMARY:
The overall purpose of this protocol is to identify subacute sepsis-associated cardiac disease in pediatric patients with cancer by CMR and evaluate the CMR findings during their follow-up. This will help inform heart failure management decision making. Evidence of dysfunction or elevated T2 values may inform adjustment of afterload reduction and beta blocker administration, and elevated ECV findings will suggest the need for increased surveillance for diastolic dysfunction.

Primary Objectives:

(Feasibility Phase) To determine the feasibility of cardiac MRI without anesthesia in the immediate post-sepsis period in children with cancer.

CMR scanning will be completed within 10 days of presentation - this will allow us to ensure that possible hemodynamic or respiratory instability and renal dysfunction has resolved prior to transport to the MRI scanner during the most acute phase of illness.

(Completion Phase) To estimate the frequency of subacute sepsis-associated cardiac disease, including myocardial inflammation and dysfunction, in the post-acute phase (within 10 days of presentation) of severe sepsis in children with cancer

DETAILED DESCRIPTION:
The primary purpose of this study is to evaluate the feasibility of obtaining cardiac MRI in pediatric patients with cancer post-septic shock which will be completed in an initial 5 patients to establish feasibility of successfully completing first study CMR within ten days of sepsis presentation without sedation.

This study will use a two-stage design. The initial stage (the feasibility phase) will evaluate the feasibility of data collection, and the second stage (the completion phase) will provide data for analysis of cardiovascular abnormalities and recovery in sepsis.

Feasibility Phase

The feasibility phase of the study will comprise the first 5 study participants. The aim of this stage is to establish feasibility of successfully completing the initial study CMR within ten days of sepsis presentation without sedation.

At completion of the feasibility phase, (first 5 participants) feasibility of data collection will be evaluated using the following stopping rule: If at least 4 of attempted 5 patient scans provide adequate available data for CMR analysis and can be completed without sedation or delay beyond the 10-day window (due to coordination or deferral due to hemodynamic instability), the study may continue to the completion phase. If fewer than 4 participants are able to complete the cardiac MRI, the study will be paused until any factors that can improve the feasibility may be identified. Data obtained during the feasibility phase will be included in analysis of CMR abnormalities.

Completion Phase

The Completion Phase will comprise approximately 20 participants in order to complete the pilot study to evaluate for abnormalities on CMR.

We estimate the feasibility phase will require up to 2 years to accrue and perform first CMR for the initial 5 patients and the completion phase will require an additional up to 18-24 months to accrue 15 additional patients who can complete CMR evaluation

ELIGIBILITY:
Inclusion Criteria:

* Between 9 and 25 years of age at time of study enrollment
* Currently receiving care for cancer at St. Jude
* Diagnosed with sepsis according to Phoenix score

Exclusion Criteria:

* Participant has been diagnosed with clinically significant left ventricular dysfunction (EF < 55%) prior to the onset of sepsis
* Participant has any condition that would, in the opinion of the investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
* Participant is pregnant
* Estimated glomerular filtration rate < 45 ml/minute/1.73m2
* Does not meet MRI safety screening criteria.

Ages: 9 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2023-05-20 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of cardiac MRI in pediatric oncology patients with sepsis | within 10 days after onset of sepsis
  The proportion of enrolled participants who have evaluable cMRI data within 10 days after onset of sepsis
Frequency of subacute sepsis-associated cardiac disease | Within 10 days of presentation
  To estimate the frequency of subacute sepsis-associated cardiac disease, including myocardial inflammation and dysfunction, in the post-acute phase (within 10 days of presentation) of severe sepsis in children with cancer

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Merlocco, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols